CLINICAL TRIAL: NCT00282659
Title: The Use of Magnesium to Improve Hemodynamics, Cholesterol, and Glucose Control: A Substudy of AdMag
Brief Title: The Use of Magnesium to Improve Blood Pressure, Cholesterol, and Glucose Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WHIT001799HI
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Hypertension; Dyslipidemia; Diabetes
Keywords: Hemodynamics; Hypertension; Dyslipidemia; Diabetes; Implantable Cardioverter Defibrillator; Blood Pressure
MeSH Terms: conditions — Coronary Artery Disease; Hypertension; Dyslipidemias; Diabetes Mellitus

INTERVENTIONS:
Drug: magnesium L-lactate

SUMMARY:
The purpose of this study is to determine if magnesium can improve blood pressure, cholesterol, and blood sugar control in patients with implantable cardioverter defibrillators (ICDs).

DETAILED DESCRIPTION:
Magnesium is the second most abundant intracellular cation and plays a vital role in many physiologic processes. It has been determined that patients with cardiovascular disease have intracellular magnesium (Mgi) deficiencies. Among the ICD registries in Europe and the United States 64% and 77% of patients also carry the diagnosis of CAD, respectively. Patients with CAD have risk factors that lead to the development and or propagation of atherosclerosis. Paramount among these risk factors are hypertension, dyslipidemia, and diabetes.

Comparison: Magnesium compared to placebo in patients with ICDs to evaluate the effect they have on cholesterol, blood pressure, and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Newly implanted ICD or recent ICD shock (within 6 months)

Exclusion Criteria:

* Inability to swallow
* A non-cardiac disease with a survival prognosis of less than 12 months
* Hypermagnesemia
* Creatinine clearance less than 30mL/min
* Lactic acidosis or systemic acidosis syndrome
* Previous intolerance to magnesium L-lactate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure, cardiac output, systemic vascular resistance, thoracic fluid content, total cholesterol, low density lipoprotein, high density lipoprotein, triglycerides, and blood glucose | at baseline, 3, and 6 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Charles M White, PharmD, Principal Investigator — University of Connecticut School of Pharmacy, Hartford Hospital Division of Drug Information
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States